CLINICAL TRIAL: NCT03921541
Title: PEACE (Pegzilarginase Effect on Arginase 1 Deficiency Clinical Endpoints): A Randomized, Double-blind, Placebo-controlled Phase 3 Study of the Efficacy and Safety of Pegzilarginase in Children and Adults With Arginase 1 Deficiency
Brief Title: Efficacy and Safety of Pegzilarginase in Patients With Arginase 1 Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aeglea Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAEB1102-300A
Record Dates: First submitted 2019-04-09; First posted 2019-04-19 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Arginase I Deficiency; Hyperargininemia
Keywords: ARG1-D
MeSH Terms: conditions — Hyperargininemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pegzilarginase (Experimental): Weekly IV infusions of pegzilarginase plus individualized disease management for 24 weeks
  Interventions: Drug: Pegzilarginase
- Placebo (Placebo Comparator): Weekly IV infusions of placebo plus individualized disease management for 24 weeks
  Interventions: Drug: Placebo
- Pegzilarginase Long Term Extension (Experimental): After completion of 24 weeks DB treatment, weekly IV infusions of pegzilarginase plus individualized disease management for an additional 150 weeks, with the option to receive treatment by SC after 8 weeks of the LTE study.
  Interventions: Drug: Pegzilarginase

INTERVENTIONS:
Drug: Pegzilarginase — Individualized disease management which includes severe protein restriction, essential amino acid supplementation and the ammonia scavengers when indicated
  Other Names: Co-ArgI-PEG; AEB1102
  Arms: Pegzilarginase; Pegzilarginase Long Term Extension
Drug: Placebo — Individualized disease management which includes severe protein restriction, essential amino acid supplementation and the ammonia scavengers when indicated
  Arms: Placebo

SUMMARY:
CAEB1102-300A is a multi-center randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of pegzilarginase in patients with ARG1-D. This study will consist of a screening period; a randomized, double-blind treatment period; a long-term extension; and a follow up visit for final safety assessments.

DETAILED DESCRIPTION:
CAEB1102-300A is a multi-center randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of pegzilarginase in patients with ARG1-D. This study will consist of a screening period; a randomized, double-blind treatment period; a long-term extension; and a follow up visit for final safety assessments.

Subjects will be randomized to treatment following completion of all screening assessments and confirmation of study eligibility in a 2:1 ratio to receive weekly IV infusions of pegzilarginase plus individualized disease management (IDM) or placebo plus IDM during the 24-week double blind treatment period. After completion of the 24-week double-blind treatment period, each subject will enter the long term, open-label extension, the first 8 weeks of which are blinded. During the long-term extension, all subjects receive pegzilarginase plus IDM. After 8 weeks of the LTE study, patients have the option to receive treatment by subcutaneous administration (SC).

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if all the following criteria apply:

1. The subject and/or parent/guardian provides written informed consent/assent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
2. A current diagnosis of ARG1 D as documented in medical records, which must include 1 of the following: elevated plasma arginine levels, a mutation analysis that results in a pathogenic variant, or reduced RBC arginase activity. For entry into this study, subjects must also fulfill the following plasma arginine criteria:

   1. The average of all measured values of plasma arginine during the screening period prior to the randomization visit (Visit 1, Study Day 1) is ≥ 250 µmol/L
   2. If a subject is re-screened, the only values that are considered for eligibility assessment are those in the current screening period
3. Subjects must be ≥ 2 years of age on the date of informed consent/assent
4. The subject must be assessable for clinically meaningful within-subject change (clinical response) on at least one component of one assessment included in the key secondary/other secondary endpoints. To be considered assessable, the subject must be able to complete the assessment, and must have a baseline deficit in at least one component as defined in the protocol
5. Have received documented confirmation from the investigator and/or dietician that the subject can maintain their diet in accordance with dietary information presented in the protocol, ie, can maintain the current level of protein consumption, including natural protein and EAA supplementation
6. Subjects receiving ammonia scavenger therapy, anti-epileptic drugs, and/or medications for spasticity (eg, baclofen) must be on a stable dose of the medication for at least 4 weeks prior to randomization and be willing to remain on a stable dose during the double-blind portion and blinded follow-up portions of the study
7. Female and male subjects may participate. Female subjects of childbearing potential must have a negative serum pregnancy test during the screening period before receiving the first dose of study treatment, and a negative urine pregnancy test on the day of the first dose, prior to the first dose. If the subject (male or female) is engaging in sexual activity that could lead to pregnancy, must be surgically sterile, postmenopausal (no menses for 12 months without an alternative medical cause or a high FSH level in the postmenopausal range in women not using hormonal contraception or hormonal replacement therapy), or must agree to use a highly effective method of birth control during the study and for a minimum of 30 days after the last study drug administration. Highly effective methods of contraception include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation; progesterone-only hormonal contraception associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); or abstinence (refraining from heterosexual intercourse during the entire period of risk associated with study treatment).

Exclusion Criteria:

1. Hyperammonemic episode (defined as an event in which a subject has an ammonia level ≥100 µM with one or more symptoms related to hyperammonemia requiring hospitalization or emergency room management) within the 6 weeks before the first dose of study drug is administered
2. Active infection requiring anti-infective therapy within 3 weeks prior to first dose
3. Known active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
4. Extreme mobility deficit, defined as either the inability to be assessed on the GFAQ or a score of 1 on the GFAQ
5. Other medical conditions or comorbidities that, in the opinion of the investigator would interfere with study compliance or data interpretation (eg, severe intellectual disability precluding required study assessments)
6. Has participated in a previous interventional study with pegzilarginase
7. Has a history of hypersensitivity to polyethylene glycol (PEG) that, in the judgment of the investigator, puts the subject at unacceptable risk for adverse events
8. Subject is being treated with botulinum toxin-containing regimens or plans to initiate such regimens during the double-blind or blinded follow-up portions of the study or received surgical or botulinum-toxin treatment for spasticity-related complications within the 16 weeks prior to the first dose of study treatment in this study
9. Is currently participating in another therapeutic clinical trial or has received any investigational agent within 30 days (or 5 half-lives whichever is longer) prior to the first dose of study treatment in this study
10. Previous liver or hematopoietic transplant procedure.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cortney Caudill, Study Director — Aeglea BioTherapeutics, Inc.
Locations (32):
- United States (17):
  - Harvey Pediatrics, Rogers, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Stanford University School of Medicine, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cohen Children's Medical Center (Northwell Health), Queens, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center Medical School at Houston, Houston, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Austria (2):
  - LKH Bregenz, Bregenz
  - Medizinische Universität Innsbruck, Innsbruck
- McGill University Health Center, Montreal, Quebec, Canada
- France (2):
  - Hôpital Necker - Enfants Malades, Paris
  - Hopital des Enfants, Talence
- Germany (2):
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
- Italy (3):
  - Fondazione MBBM, Monza
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- United Kingdom (5):
  - Birmingham Children's Hospital, Birmingham
  - University Hospital of Wales, Cardiff
  - Great Ormond Street Hospital for Children, London
  - Willink Biochemical Genetics Unit, Manchester
  - Salford Royal, Salford

REFERENCES:
- [Derived] Russo RS, Gasperini S, Bubb G, Neuman L, Sloan LS, Diaz GA, Enns GM; PEACE Investigators. Efficacy and safety of pegzilarginase in arginase 1 deficiency (PEACE): a phase 3, randomized, double-blind, placebo-controlled, multi-centre trial. EClinicalMedicine. 2024 Jan 12;68:102405. doi: 10.1016/j.eclinm.2023.102405. eCollection 2024 Feb. PMID 38292042

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegzilarginase: Weekly IV infusions of pegzilarginase plus individualized disease management for 24 weeks
  After completion of the 24-week double-blind treatment period, each subject entered the long term, open-label extension where all subjects received weekly SC or IV pegzilarginase plus individualized disease management
- Placebo: Weekly IV infusions of placebo plus individualized disease management for 24 weeks
  After completion of the 24-week double-blind treatment period, each subject entered the long term, open-label extension where all subjects received weekly SC or IV pegzilarginase plus individualized disease management
Period: Double Blind Treatment Period
Arm/Group | Pegzilarginase | Placebo
Started | 21 | 11
Completed | 20 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Long Term Extension
Arm/Group | Pegzilarginase | Placebo
Started | 20 | 11
Completed | 20 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegzilarginase | Placebo | Total
Number analyzed (Participants) | 21 | 11 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 9 | 29
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (6.16) | 12.9 (6.77) | 10.7 (6.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 12 | 7 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 10 | 4 | 14
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 7 | 1 | 8
Age at Diagnosis [Mean (Standard Deviation); unit: years] | 2.8 (4.06) | 4.2 (3.07) | 3.3 (3.75)
GMFCS Level [Count of Participants; unit: Participants] — The GMFCS assigns gross motor function capabilities based on movements such as sitting, walking, and use of mobility devices with 5 categories ranging from I (most functional) to V (transported in wheelchair in all settings)
  Participants
    I | 9 | 5 | 14
    II | 9 | 4 | 13
    III | 0 | 0 | 0
    IV | 3 | 2 | 5
    V | 0 | 0 | 0
Level of Spasticity [Count of Participants; unit: Participants]
  None | 8 | 3 | 11
  Mild | 7 | 2 | 9
  Moderate | 5 | 4 | 9
  Severe | 1 | 2 | 3
Historical arginine level [Mean (Standard Deviation); unit: micromolar] — Population: Data not available for 2 subjects in pegzilarginase group.
  micromolar
    number analyzed (Participants) | 19 | 11 | 30
    (all) | 409.4 (114.83) | 476.1 (124.09) | 433.9 (120.68)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Arginine Concentration After 24 Weeks of Treatment
Description: The primary analysis will test the change in the level of plasma arginine between baseline and completion of week 24 assessments. It will compare the change from baseline in plasma arginine between participants treated with pegzilarginase and those treated with placebo.
Time Frame: Baseline through Week 24
Population: Full Analysis Set - all subjects who are randomized and who receive at least 1 dose of blinded study treatment
Measure: Geometric Mean (Standard Deviation); unit: micromolar
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 21 | 11
micromolar | 0.244 (1.635) | 0.918 (1.371)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: Mean Change From Baseline in the Mobility Assessments of the Key Secondary Outcome Measure of the 2 Minute Walk Test
Description: The Key Secondary outcome measure is the mean change from baseline in the 2 Minute Walk Test.
Time Frame: Baseline through Week 24
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 19 | 10
meters | 7.3 (30.64) | 2.7 (19.66)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p = 0.5961, Mixed Models Analysis

3. Secondary Outcome: Mean Change From Baseline in the Mobility Assessments of the Key Secondary Outcome Measure of GMFM-E
Description: The Key Secondary outcome measure is the mean change from baseline in GMFM-E
  The Gross Motor Function Measure (GMFM) utilize a 4-point scoring system for each item across dimensions A-E. GMFM-E assesses walking, running, and jumping. The minimum score for GMFM-E is 0; the maximum score is 72, with a higher score representing better gross motor function
Time Frame: Baseline through Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 20 | 11
score on a scale | 4.2 (7.69) | -0.4 (6.20)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p = 0.1087, Mixed Models Analysis

4. Secondary Outcome: Proportion of Participants With Plasma Arginine Levels Below Target Guidance
Description: Proportion of participants with plasma arginine levels below 200umol/L (target level set in disease management guidelines) after 24 weeks of treatment.
Time Frame: Baseline and week 24
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 21 | 11
Participants | 19 | 0
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact

5. Secondary Outcome: Proportion of Participants With Plasma Arginine Levels in Normal Range
Description: Proportion of participants with plasma arginine levels between 40 - 115 umol/L (normal range for plasma arginine) after 24 weeks.
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 21 | 11
Participants | 19 | 0
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact

6. Secondary Outcome: Change in Ornithine
Description: This analysis will measure the change from baseline in the level of ornithine after 24 weeks of treatment.
Time Frame: Baseline and week 24
Measure: Geometric Least Squares Mean (Standard Error); unit: micromolar
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 15 | 10
micromolar | 1.941 (1.087) | 0.938 (1.107)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

7. Secondary Outcome: Change in Guanidino Compound-ARGA
Description: This analysis will measure the change from baseline in the level of ARGA after 24 weeks of treatment.
Time Frame: Baseline to week 24
Measure: Geometric Least Squares Mean (Standard Error); unit: micromolar
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 21 | 11
micromolar | 0.306 (1.099) | 1.003 (1.141)

8. Secondary Outcome: Change in Guanidino Compound - GAA
Description: This analysis will measure the change from baseline in the level of GAA compound after 24 weeks of treatment.
Time Frame: Baseline to week 24
Measure: Geometric Least Squares Mean (Standard Error); unit: micromolar
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 21 | 11
micromolar | 0.481 (1.111) | 1.030 (1.157)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p = 0.0003, Mixed Models Analysis

9. Secondary Outcome: Change in Guanidino Compound - GVA
Description: This analysis will measure the change from baseline in the level of GVA compound after 24 weeks of treatment.
Time Frame: Baseline to week 24
Measure: Geometric Least Squares Mean (Standard Error); unit: micromolar
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 21 | 11
micromolar | 0.290 (1.108) | 0.916 (1.153)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

10. Secondary Outcome: Change in Guanidino Compound - NAArg
Description: This analysis will measure the change from baseline in the level of NAArg compound after 24 weeks of treatment.
Time Frame: Baseline to week 24
Measure: Geometric Least Squares Mean (Standard Error); unit: micromolar
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 21 | 11
micromolar | 0.289 (1.140) | 0.956 (1.200)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

11. Secondary Outcome: Mean Change From Baseline at Week 24 in Other Aspects of Mobility Assessed by GMFM-D
Description: To compare pegzilarginase with placebo with respect to other aspects of mobility.
  The Gross Motor Function Measure (GMFM) utilize a 4-point scoring system for each item across dimensions A-E. GMFM-D assesses tasks related to standing. The minimum score for GMFM-D is 0; the maximum score is 39 with a higher score representing better gross motor function
Time Frame: Baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 20 | 11
score on a scale | 2.7 (3.88) | 0.4 (0.97)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p = 0.0208, Mixed Models Analysis

12. Secondary Outcome: Mean Change From Baseline at Week 24 in Other Aspects of Mobility Assessed by the Functional Mobility Scale (FMS)
Description: To compare pegzilarginase with placebo with respect to other aspects of mobility utilizing the FMS-5 Score.
  The functional mobility scale (FMS) is a 6-point scale from Level 1 (uses wheelchair, stroller, scooter, shopping cart, wagon, or is carried OR walks for exercise only with highly specialized/ supportive walker OR does limited stepping with substantial support/assistance from another person) to Level 6 (independent walking and running on all surfaces without assistive devices or help from another person) that assesses the need for assistive devices for walks of 3 different lengths: 5 meters, 50 meters, and 500 meters.
Time Frame: Baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 20 | 11
score on a scale | 0.1 (0.39) | -0.1 (0.70)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p = 0.4434, Mixed Models Analysis

13. Secondary Outcome: Mean Change From Baseline at Week 24 in Other Aspects of Mobility Assessed by the Functional Mobility Scale (FMS)
Description: To compare pegzilarginase with placebo with respect to other aspects of mobility utilizing the FMS-50 Score.
  The functional mobility scale (FMS) is a 6-point scale from Level 1 (uses wheelchair, stroller, scooter, shopping cart, wagon, or is carried OR walks for exercise only with highly specialized/ supportive walker OR does limited stepping with substantial support/assistance from another person) to Level 6 (independent walking and running on all surfaces without assistive devices or help from another person) that assesses the need for assistive devices for walks of 3 different lengths: 5 meters, 50 meters, and 500 meters.
Time Frame: Baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 19 | 11
score on a scale | 0.2 (0.42) | 0.1 (0.83)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p = 0.5301, Mixed Models Analysis

14. Secondary Outcome: Mean Change From Baseline at Week 24 in Other Aspects of Mobility Assessed by the Functional Mobility Scale (FMS)
Description: To compare pegzilarginase with placebo with respect to other aspects of mobility utilizing the FMS-500 Score.
  The functional mobility scale (FMS) is a 6-point scale from Level 1 (uses wheelchair, stroller, scooter, shopping cart, wagon, or is carried OR walks for exercise only with highly specialized/ supportive walker OR does limited stepping with substantial support/assistance from another person) to Level 6 (independent walking and running on all surfaces without assistive devices or help from another person) that assesses the need for assistive devices for walks of 3 different lengths: 5 meters, 50 meters, and 500 meters.
Time Frame: Baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 18 | 11
score on a scale | 0.1 (0.24) | 0.2 (0.40)
Statistical Analysis 1: Comparison: Pegzilarginase vs Placebo; Test type: Superiority; p = 0.2515, Mixed Models Analysis

15. Secondary Outcome: Mean Change From Baseline at Week 24 in Other Aspects of Mobility Assessed by the Gillette Functional Assessment Questionnaire (GFAQ)
Description: To compare pegzilarginase with placebo with respect to other aspects of mobility.
  The Gillette Functional Assessment Questionnaire (GFAQ) is a parent/caregiver assessment consisting of a single question describing a child's ability to walk using a 10-point scale from Level 1 (cannot take any steps at all) to Level 10 (walks, runs, and climbs on uneven terrain and does stairs without difficulty or assistance; is typically able to keep up with peers).
Time Frame: Baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 20 | 11
score on a scale | 0.1 (0.79) | -0.3 (0.90)

16. Secondary Outcome: Mean Change From Baseline at Week 24 in Adaptive Behavior Assessed Using the Vineland Adaptive Behavior Scales (VABS)-II
Description: To compare pegzilarginase with placebo with respect to adaptive behavior.
  The Vineland Adaptive Behavior Scales (VABS-II) is a scale designed to measure adaptive behavior of individuals from birth to age 90 years. The VABS-II contains 4 domains: communication, daily living skills, socialization, and motor skills. The domains are made up of 11 subdomains in which the scores are added to form the domain composite scores. The 4 domain composite scores then combine to form the adaptive behavior composite for those individuals aged birth to 6 years 11 months. Three domain composite scores (communication, daily living skills, and socialization) combine to form the adaptive behavior composite for those ages 7 through 90 years. The VABS-II scoring system describes adequate adaptive behavior by subdomain as 13 to 17 and 86 to 114 for the composite score, with higher scores indicating better adaptive functioning.
Time Frame: Baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 18 | 10
score on a scale | 1.4 (16.54) | -1.6 (8.78)

17. Secondary Outcome: Evaluate Safety of Pegzilarginase
Description: Number of participants developing treatment related adverse events.
Time Frame: Reporting will be from signing consent through follow-up (Baseline to Week 24)
Measure: Count of Participants; unit: Participants
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 21 | 11
Participants | 18 | 11

18. Secondary Outcome: Evaluate Immunogenicity of Pegzilarginase
Description: The proportion of participants who develop (ADA) anti-drug antibodies to pegzilarginase will be measured over the period of the clinical trial.
Time Frame: Baseline to week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegzilarginase | Placebo
Number analyzed (Participants) | 21 | 11
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Baseline to 24 weeks
Arm/Group | Pegzilarginase | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 4/21 | 4/11
Other Adverse Events (participants affected / at risk) | 18/21 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegzilarginase (N=21) | Placebo (N=11)
Hyperammonaemia (Metabolism and nutrition disorders) | 2 | 3
Hyperammonaemic encephalopathy (Metabolism and nutrition disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegzilarginase (N=21) | Placebo (N=11)
Abdominal Pain (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 5 | 3
Pyrexia (General disorders) | 4 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Ammonia increased (Investigations) | 3 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood potassium decreased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1
Generalized anxiety disorder (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT03921541/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT03921541/SAP_001.pdf